CLINICAL TRIAL: NCT04235816
Title: Evaluation of the Impact on Childhood Mortality of Azithromycin Plus Intermittent Preventive Treatment Administered Through the Expanded Program on Immunization in Sierra Leone
Brief Title: Improving Care Through Azithromycin Research for Infants in Africa
Acronym: ICARIA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Barcelona Institute for Global Health (Other)
Collaborators: University of Sierra Leone (Other); Bill and Melinda Gates Foundation (Other); Ministry of Health and Sanitation, Sierra Leone (Other Government); La Caixa Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ICARIA; OPP1196642 (Other Grant/Funding Number: Bill & Melinda Gates Foundation)
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Child Mortality
Keywords: Infant; U5; Azithromycin; Intermittent preventive treatment for infants; Expanded Program on Immunization; Malaria; Sulphadoxine-pyrimethamine
MeSH Terms: conditions — Malaria | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: 2-arm individually randomized placebo-controlled clinical trial of AZi administration in young children from Sierra Leone.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple: (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (Active Comparator): AZi at DTP-1 visit at 6 weeks of age, AZi (plus IPTi) at measles visit at 9 months of age and AZi (plus IPTi) at measles booster visit at 15 months of age.
  Interventions: Drug: Azithromycin
- Group 2 (Placebo Comparator): Placebo at DTP-1 visit at 6 weeks of age, placebo (plus IPTi) at measles visit at 9 months of age and placebo (plus IPTi) at measles booster visit at 15 months of age.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — Administration of azithromycin during the first 15 months of life through the Expanded Program on Immunisation
  Other Names: AZi; Sumamed
  Arms: Group 1
Drug: Placebo — Administration of placebo during the first 15 months of life through the Expanded Program on Immunisation
  Arms: Group 2

SUMMARY:
Infectious diseases are among the most common causes of mortality in the over 2.5 million children under 5 years of age (U5) who died in 2018 in sub-Saharan Africa (SSA). New approaches to treatment and prevention of these diseases are needed to increase child survival. Sierra Leone has one of the highest rates of under-five child mortality in the world. It is estimated that 32,000 children die each year, the leading causes being neonatal conditions, malaria, pneumonia and diarrhea. In Sierra Leone, the available information on malaria indicates that it accounts for 38% of deaths among under-five children. Reducing the prevalence and impact of the disease among the general population is a major priority of the Ministry of Health and Sanitation (MoHS) of Sierra Leone .

Intermittent Preventative Treatment in infants (IPTi) - the administration of a full course antimalarial treatment to infants at individual timepoints regardless of infection status- has been shown to reduce clinical malaria and anemia in infants in the first year of life . When delivered alongside the Expanded Program on Immunization (EPI), IPTi with Sulphadoxine-pyrimethamine (SP) is a highly cost-effective intervention. . Sierra Leone is currently the only country that implements nationwide the World Health Organization's (WHO) IPTi guideline, which is administered within the first year of life. However, its benefit when expanded into the second year of life remains unknown. Taking the advantage of the inclusion in the EPI program of a booster dose of measles vaccine at 15 months of age, the ICARIA trial will also assess the efficacy of adding a dose of IPTi-SP at this age.

Recent studies show that azithromycin (AZi) - a macrolide antibiotic with some antimalarial effect- is associated with a significant reduction in childhood mortality when used in mass drug administration (MDA) for trachoma elimination in areas of sub-Saharan Africa (SSA) with child mortality rates far beyond Sustainable Development Goals , . However, despite the potential benefit of the intervention several fundamental scientific questions need to be answered before it can be recommended for large-scale implementation.

DETAILED DESCRIPTION:
In order to generate the conclusive evidence needed to inform policy and accelerate the implementation of this intervention, we propose to carry out a large-scale clinical trial on the impact on all-cause mortality up to 18 months of age of AZi administration through EPI. The potential development of antibiotic and SP resistance, AZi and SP interactions with routine immunizations, as well as the safety and the impact on the health system will be all assessed in the ICARIA trial.

To provide the evidence needed to inform policy and practice and to accelerate the implementation of this intervention, a large-scale clinical trial on the impact on all-cause mortality up to 18 months of age of AZi administration through the World Health Organisation Expanded Program on Immunisation (EPI) will be carried out in Sierra Leone. The clinical trial will be individually randomised, placebo-controlled with a factorial design whereby AZi will be administered alongside routine preventive health interventions of the EPI, such as immunisations and Intermittent Preventive Treatment in infants (IPTi), which is recommended by the WHO for malaria prevention in this age group. The potential development of antibiotic resistance, the interactions with routine immunisations, the safety and the impact on the health system of AZi administration will be all assessed in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Parents/guardians have signed the informed consent
* Permanent residence in the study area-health facility catchment area
* Without known allergies to or contraindications to macrolides
* Without known allergies to or contraindications to SP
* Agreement to complete the EPI scheme at the recruitment health facility
* Parents/guardians agree to participate

Exclusion Criteria:

* Residence outside the study area or planning to move out in the following 12 months from enrolment
* Known history of allergy or contraindications to macrolides and/or SP
* Known history of allergy or contraindications to SP
* With signs of any acute illness at the time of recruitment
* Participating in other intervention studies

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20560 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2025-09-11 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
The rate of all-cause mortality | 18 months of age
  all-cause mortality rate at 18 months of age

SECONDARY OUTCOMES:
The cause-specific mortality rate | 18 months of age
  Cause-specific mortality rate at 18 months of age
Malaria related mortality | 18 month of age
  Malaria related mortality at 18 months of age
Incidence of all-cause hospital admissions | Through study completion, 36 months
  Incidence of all-cause hospital admissions
Incidence of all-cause outpatient attendances | Through study completion, 36 months
  Incidence of all-cause outpatient attendances at the health facilities
Incidence of confirmed (RDT positive) malaria hospital admissions | Through study completion, 36 months
  Incidence of confirmed (RDT positive) malaria hospital admissions at all health facilities
Incidence of confirmed (blood smear positive/RDT positive) malaria hospital admissions | Through study completion, 36 months
  Incidence of confirmed (blood smear positive/RDT positive) malaria hospital admissions at all health facilities
Frequency and severity of drug adverse reactions | Through study completion, 36 months
  Frequency and severity of drug adverse reactions throughout the trial
Prevalence of macrolide resistance in nasopharyngeal isolates | Through study completion, 36 months
  Prevalence of macrolide resistance in nasopharyngeal isolates
Prevalence of macrolide resistance in the gut bacteria | Through study completion, 36 months
  Prevalence of macrolide resistance in the gut bacteria
Proportion of children with protective antibody responses to specific routine EPI immunizations (measles and yellow fever) | Through study completion, 36 months
  Proportion of children with protective antibody responses to specific routine EPI

CONTACTS AND LOCATIONS:
Overall Officials: Clara Menendez, MD, PhD, Principal Investigator — Barcelona Institute for Global Health
Locations (1):
- College of Medicine and Allied Health Sciences, Freetown, Sierra Leone

REFERENCES:
- [Derived] Chen H, Owusu-Kyei K, Fombah AE, Williams J, Garcia-Fernandez C, Rovira-Vallbona E, Bofill A, Quinto L, Figueroa-Romero A, Mac-Abdul F, Samai M, Mayor A, Menendez C. Prevalence of Molecular Markers of Resistance to Antimalarial Drugs Three Years After Perennial Malaria Chemoprevention in Sierra Leone. Gates Open Res. 2025 Oct 8;9:81. doi: 10.12688/gatesopenres.16367.1. eCollection 2025. PMID 41080970
- [Derived] Owusu-Kyei K, Chen H, Chileshe M, Quinto L, Sibley M, Figueroa-Romero A, Llach M, Ramirez M, Bofill A, Samai M, Menendez C; ICARIA Trial Team. Impact of oral azithromycin and intermittent preventive treatment with sulfadoxine-pyrimethamine regimen on child mortality in Sierra Leone: trial protocol for a randomised, two-arm, double-blinded, placebo-controlled clinical trial (ICARIA). Trials. 2024 Sep 27;25(1):626. doi: 10.1186/s13063-024-08443-9. PMID 39334260